CLINICAL TRIAL: NCT00426699
Title: Urinary Excretion of Enteroviruses From Children With a Presumed Enteroviral Infection
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Andreas Pasch, Department of Nephrology and Hypertension, Inselspital, University Hospital Bern
Other Study IDs: BE002
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Enterovirus Infections
Keywords: enterovirus; meningitis; sepsis; myocarditis; kidney; urine; glomerulonephritis
MeSH Terms: conditions — Enterovirus Infections; Meningitis; Sepsis; Myocarditis; Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Enteroviruses can infect most human organ systems, especially the heart, nervous system and pancreas. Whether Enteroviruses can also affect the kidneys is not known yet. Therefore we will analyze urine of children with a suspected enteroviral infection for enteroviruses and signs of kidney infection.

DETAILED DESCRIPTION:
Enteroviruses have been shown to cause mesangioproliferation and glomerulonephritis in mice (especially coxsackievirus B4). In some cases, large amounts of IgA are deposited in the mesangium, resembling human IgA-nephropathy. In humans, case reports indicate the propensity of certain enteroviruses to cause kidney infections.

Our project aims to analyze urine of children with suspected enteroviral infections (e.g. meningitis, myocarditis, sepsis of the newborn etc.) to identify cases suspicious of concomitant enteroviral kidney affection. To achieve this aim, enterovirus-PCRs will be performed and microhematuria searched for.

ELIGIBILITY:
Inclusion Criteria:

* children, suspected of suffering from an enteroviral infection

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children age 0-16
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pasch, MD, Principal Investigator — University of Bern
Locations (1):
- Dept. Nephrology & Hypertension, Univ. Hospital Bern, Bern, Canton of Bern, Switzerland